CLINICAL TRIAL: NCT00921596
Title: Cardiac Operation Under Totally Endoscope and Cardiopulmonary Bypass, a Single Center's Experience
Brief Title: Cardiac Operation Under Totally Endoscope and Cardiopulmonary Bypass (CPB)
Acronym: CPB
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Shiqiang Yu, Xijing Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: xinzangwaike0003
Record Dates: First submitted 2009-06-12; First posted 2009-06-16 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Congenital Heart Defects; Heart Valve Diseases
Keywords: Surgical Procedures, Cardiac; Minimally Invasive Surgical Procedures; Thoracoscopes; Cardiopulmonary Bypass
MeSH Terms: conditions — Heart Defects, Congenital; Heart Valve Diseases | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Totally endoscopic cardiac operation (Other): Patients with cardiac diseases undergo cardiac operations with totally endoscopic and cardiopulmonary bypass
  Interventions: Procedure: cardiac operation with totally endoscopic method

INTERVENTIONS:
Procedure: cardiac operation with totally endoscopic method — Cardiac operations are performed with three keyholes in the right chest wall. Video images are obtained by digital thoracoscope through one hole. Intracardiac lesions are accessed with surgical instruments and repaired through the other two holes. Cardiopulmonary bypass is set up with femoral cannulations. Moderate system hypothermic is applied for the operation. Cardiac arrest is achieved with ascending aorta clamp and cardioplegia solution delivery through aortic root cannulation. After the intracardiac lesions are repaired, aortic clamp is removed, and the heart is reperfused to restore its spontaneous rhythm. After the patients are rewarmed to normal temperature, CPB is discontinued. Femoral cannulations are removed, and surgical wounds are closed.
  Other Names: thoracoscopic cardiac surgery

SUMMARY:
Conventional cardiac operations are performed with median sternotomy, which is related to great wound, morbidities, longer duration in hospital and most significantly, cosmetic problems. The investigators invested a new minimally invasive cardiac operation method totally under video-endoscope and peripheral cardiopulmonary bypass. The investigators' hypothesis is that this new minimally method could provide better cosmetic effects to the patients, and also relate to shorter postoperative hospital stay and better recovery.

ELIGIBILITY:
Inclusion Criteria:

* congenital heart defects or heart valve diseases require surgical correction

Exclusion Criteria:

* Body weight < 10kg
* committed with complex congenital heart defect
* anticipated to perform aortic valve repair or replacement
* anticipated to perform aorta repair or replacement
* committed with Femoral vessel diseases unable to perform femoral cannulation
* refuse to perform totally thoracoscope minimally invasive surgery

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2000-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | one year

SECONDARY OUTCOMES:
all cause morbidity | one year

CONTACTS AND LOCATIONS:
Overall Officials: Dinghua Yi, MD, Study Chair — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shannxi, China